CLINICAL TRIAL: NCT02949141
Title: Diagnostic Use of Lung Ultrasound Compared to Chest X-Ray for Suspected Pneumonia in Nepal
Brief Title: Diagnostic Use of Lung Ultrasound for Suspected Pneumonia in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patan Academy of Health Sciences (Other)
Collaborators: Vanderbilt University (Other); Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Darlene Rose House, Assistant Professor of Clinical Emergency Medicine and Pediatrics, Patan Academy of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pahs
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound (Experimental): All patients will initially get an ultrasound (interpreted by emergency department physician) followed by chest x-ray (read by independent radiologist) and computed tomography (read by radiologist)
  Interventions: Device: Lung Ultrasound; Device: Chest X-ray; Device: Chest Computed Tomography (CT)

INTERVENTIONS:
Device: Lung Ultrasound — All patients will receive lung ultrasound, chest x-ray and computed tomography
Device: Chest X-ray — All patients will receive chest x-ray as per usual care for evaluation for pneumonia
Device: Chest Computed Tomography (CT) — All enrolled patients will receive a CT scan as the gold standard for diagnosing pneumonia

SUMMARY:
This study is designed to evaluate the use of lung ultrasound compared to chest x-ray to diagnose pneumonia in Nepal. Given the ease, portability, and relative ease of teaching ultrasound, this would be potential technology available for many clinicians throughout Nepal to use for adult and pediatric patients presenting with suspected pneumonia. This would be especially useful in remote areas where clinicians have limited access to x-rays. Despite its utility, use of ultrasound to diagnose pneumonia in resource-limited settings like Nepal has not yet been studied. Therefore, this study is designed as a prospective, clinical diagnostic study to evaluate patients presenting with suspected pneumonia using diagnostic imaging of beside ultrasound compared with chest x-ray using computed tomography as the gold standard for diagnosis of pneumonia.

DETAILED DESCRIPTION:
Study Design: A prospective, convenience sample of participants presenting with suspected pneumonia when trained ultrasound investigator is present in the Patan Hospital Emergency Department will be performed in Patan, Nepal. This study will be done in partnership with Patan Hospital Emergency Department and with the approval of Nepal Health Research Council and Patan Hospital's ethical review committee.

Study Setting: Located in the Kathmandu valley, Patan Hospital is a large urban hospital with 35-bed Emergency Department that sees approximately 32,000 patients per year.

Study Protocol:

Prior to the enrolling patients, investigators in the Emergency Department will save lung ultrasound exams and interpret the exams. These exams will then be independently reviewed by an ultrasonographer to ensure adequate skill in lung ultrasonography. A kappa analysis of these scans will be performed. If kappa <0.6, we will review lung ultrasound with these investigators and repeat above evaluation until kappa of 0.6 is achieved.

For participants meeting inclusion criteria, consent will be obtained from the participant. Consent will include explanation of use of bedside ultrasound and chest CT scan for diagnosis of their condition. This consent will also include explanation of risks and benefits in Nepali. These examinations will be provided free of charge to the participant.

The investigator will record patient demographics, symptoms, lung exam findings, and pre-test probability of pneumonia (low, intermediate, high) on the data form.

After initial clinical evaluation, a bedside lung ultrasound will be performed. A Sonosite M Turbo (Fujifilm Sonosite, Inc.) ultrasound machine will be used. The ultrasound examination will include ten views, two anterior views, two lateral views (one including the costophrenic angle), and one posterior view on both chest walls. The investigator will then record findings and diagnosis on the data entry form along with their post-test probability of pneumonia (low, intermediate, high).

Participants will get a chest x-ray as a part of the standard evaluation. These readings will be recorded on the data sheet. Participants will then undergo a chest computed tomography (CT), as the diagnostic standard to evaluate for pneumonia. The chest x-ray and chest CT will be read by a radiologist. The radiologist will be blinded to the results of the previous studies. The reading and diagnosis according to CT will be recorded on the data form.

Statistical Analysis

The performance of ultrasound for diagnosis of pneumonia will be expressed as sensitivity, specificity, and likelihood ratios. Since the sensitivity of ultrasound is estimated around 90%, in order to detect a 20% difference based on a CXR sensitivity of 70%, 62 patients will be needed. McNemar's test will be used to evaluate any statistical difference in sensitivity between CXR and US.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Emergency Department at Patan Hospital age 18 or older with suspected signs of pneumonia with at least three of the following: temperature greater than 38 or history of fever, cough, dyspnea, heart rate higher than 100 beats per minute, or oxygen saturation lower than 92%.

Exclusion Criteria:

* Children will be excluded from the study. Also, ultrasound studies completed by physicians not trained in lung ultrasound will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bharat Yadav, MD, Study Chair — Chair of Department of Emergency Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cortellaro F, Colombo S, Coen D, Duca PG. Lung ultrasound is an accurate diagnostic tool for the diagnosis of pneumonia in the emergency department. Emerg Med J. 2012 Jan;29(1):19-23. doi: 10.1136/emj.2010.101584. Epub 2010 Oct 28. PMID 21030550
- [Result] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Result] Bourcier JE, Paquet J, Seinger M, Gallard E, Redonnet JP, Cheddadi F, Garnier D, Bourgeois JM, Geeraerts T. Performance comparison of lung ultrasound and chest x-ray for the diagnosis of pneumonia in the ED. Am J Emerg Med. 2014 Feb;32(2):115-8. doi: 10.1016/j.ajem.2013.10.003. Epub 2013 Oct 9. PMID 24184011
- [Result] Hagaman JT, Rouan GW, Shipley RT, Panos RJ. Admission chest radiograph lacks sensitivity in the diagnosis of community-acquired pneumonia. Am J Med Sci. 2009 Apr;337(4):236-40. doi: 10.1097/MAJ.0b013e31818ad805. PMID 19365166
- [Result] Liu XL, Lian R, Tao YK, Gu CD, Zhang GQ. Lung ultrasonography: an effective way to diagnose community-acquired pneumonia. Emerg Med J. 2015 Jun;32(6):433-8. doi: 10.1136/emermed-2013-203039. Epub 2014 Aug 20. PMID 25142033
- [Result] Reissig A, Copetti R, Mathis G, Mempel C, Schuler A, Zechner P, Aliberti S, Neumann R, Kroegel C, Hoyer H. Lung ultrasound in the diagnosis and follow-up of community-acquired pneumonia: a prospective, multicenter, diagnostic accuracy study. Chest. 2012 Oct;142(4):965-972. doi: 10.1378/chest.12-0364. PMID 22700780
- [Result] Reissig A, Gramegna A, Aliberti S. The role of lung ultrasound in the diagnosis and follow-up of community-acquired pneumonia. Eur J Intern Med. 2012 Jul;23(5):391-7. doi: 10.1016/j.ejim.2012.01.003. Epub 2012 Feb 21. PMID 22726366
- [Result] Syrjala H, Broas M, Suramo I, Ojala A, Lahde S. High-resolution computed tomography for the diagnosis of community-acquired pneumonia. Clin Infect Dis. 1998 Aug;27(2):358-63. doi: 10.1086/514675. PMID 9709887
- [Derived] Amatya Y, Rupp J, Russell FM, Saunders J, Bales B, House DR. Diagnostic use of lung ultrasound compared to chest radiograph for suspected pneumonia in a resource-limited setting. Int J Emerg Med. 2018 Mar 12;11(1):8. doi: 10.1186/s12245-018-0170-2. PMID 29527652

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients eligible for the study were included and received all three imaging modalities.
Groups:
- All Participants: All patients will initially get an ultrasound (interpreted by emergency department physician) followed by chest x-ray (read by independent radiologist) and computed tomography (read by radiologist)
  Lung Ultrasound: All patients will receive lung ultrasound, chest x-ray and computed tomography.
Period: Overall Study
Arm/Group | All Participants
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ultrasound: All patients will initially get an ultrasound (interpreted by emergency department physician) followed by chest x-ray (read by independent radiologist) and computed tomography (read by radiologist)
  Lung Ultrasound: All patients will receive lung ultrasound, chest x-ray and computed tomography.
  No adverse events were recorded.
Arm/Group | Ultrasound
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Nepal | 62

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis of Pneumonia
Description: Sensitivity and specificity of ultrasound compared to chest x-ray for the diagnosis of pneumonia using Chest CT as the gold standard for diagnosis.
Time Frame: 9 months
Population: 62
Measure: Count of Participants; unit: Participants
Groups:
- Ultrasound: Ultrasound Diagnosis of pneumonia compared to CT (Gold Standard)
- Chest X-Ray: Chest x-ray diagnosis of pneumonia compared to CT
Arm/Group | Ultrasound | Chest X-Ray
Number analyzed (Participants) | 62 | 62
Participants
  US (or CXR) and CT positive pneumonia | 40 | 32
  US (or CXR) negative, CT positive | 4 | 12
  US (or CXR) positive, CT negative | 7 | 9
  US (or CXR) negative, CT negative | 11 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during hospital stay.
Description: No adverse events
Groups:
- Ultrasound: Lung Ultrasound evaluation for pneumonia.
  All patients will receive lung ultrasound, chest x-ray and computed tomography.
  No adverse events were recorded.
- Chest X-ray: Chest x-ray for evaluation of pneumonia.
- Chest Ct: Following US and CXR, all patients received a Chest CT as the gold standard for diagnosis of pneumonia.
Arm/Group | Ultrasound | Chest X-ray | Chest Ct
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT02949141/Prot_SAP_002.pdf
  • Informed Consent Form (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT02949141/ICF_003.pdf